CLINICAL TRIAL: NCT06094972
Title: The Effectiveness of A-CRA in Compulsory Institutional Care for Youth - an Independent Randomized Controlled Trial
Brief Title: The Effectiveness of A-CRA in Compulsory Institutional Care for Youth
Acronym: A-CRA at SiS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tobias Lundgren, PhD, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-06079-01
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Substance Use Disorders; Criminal Behavior
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + A-CRA (Experimental): TAU: Interventions and treatments usually offered and delivered in institutional care. See below for examples.
  12-14 weekly sessions of A-CRA, a behavioral treatment for youth suffering from substance use disorder and co-occurring problems. Treatment consists of 18 procedures that aim to reduce problematic behaviors and increase constructive behaviors. Examples of procedures are functional analysis of substance use behavior, functional analysis of prosocial behavior, increasing prosocial activities, drink/drug refusal, relapse prevention, anger management and caregiver sessions. Procedures are combined and tailored to meet youth individual goals and needs.
  Interventions: Behavioral: Adolescent Community Reinforcement Approach, A-CRA
- TAU (Active Comparator): Standard care is defined as the interventions and treatments adolescents are usually offered and undergo in institutional care. These are Motivational Interviewing, MI, Cognitive Behavioral Therapy, CBT, Aggression Replacement Therapy, ART or Acceptance and Commitment Therapy, ACT. This will be further specified and registered in the initial phase of the study, in collaboration with SiS.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Adolescent Community Reinforcement Approach, A-CRA — A-CRA consists of eighteen treatment modules/procedures that is delivered in weekly sessions over 12-14 weeks. The overarching goal is to decrease substance use behaviours and other related, problematic behaviours such as acting out when experiencing anger, and to increase prosocial and sober behaviours, relationships and activities. The procedures are: 1) Introduction to A-CRA/treatment agreement, 2) Happiness scale and treatment goals, 3) Homework, 4) Systematic encouragement, 5) Functional analysis of substance use behaviour, 6) Functional analysis of prosocial/sober behaviour, 7) Increasing prosocial activities, 8) Drink/drug refusal, 9) Relapse prevention, 10) Sobriety sampling, 11) Communication skills, 12) Problem-solving, 13) Caregiver sessions, 14) Relationship skills, 15) Couple relationship skills, 16) Job-seeking skills, 17) Anger management, 18) Medication adherence and monitoring. Youths' individual goals and problems guide treatment planning.
  Arms: TAU + A-CRA
Behavioral: TAU — Standard care is defined as the interventions and treatments adolescents are usually offered and undergo in institutional care in Sweden. These are Motivational Interviewing, MI, Cognitive Behavioral Therapy, CBT, Aggression Replacement Therapy, ART or Acceptance and Commitment Therapy, ACT and PULS, a program for reducing violence and criminal behavior. Also, individually tailored interventions will be included, such as counselling or other psychological interventions. TAU will be thoroughly registered during the study since the sites in the trial differs slightly in what they offer.
  Arms: TAU

SUMMARY:
Youth with substance use disorder (SUD) and socially disruptive behaviour (such as criminality) who are placed in compulsory institutional care are at high risk of continuing a destructive lifestyle into adulthood. There is a pressing need for effective treatment for this group, yet studies are scarce. The empirically supported SUD treatment Adolescent Community Reinforcement Approach, A-CRA, promotes long-term abstinence, increases social stability and decreases co-morbid psychiatric problems for youth ages 12-25. A-CRA is proven to be one of the most effective SUD treatments for youth but has only been evaluated in outpatient care. Given A-CRA's promising results for youth in vulnerable living situations, it is a reasonable treatment to adjust and evaluate in compulsory care. The main objectives are to evaluate the effectiveness of A-CRA, the short- and long-term effects on social-, emotional- and problem behavior and substance use, for youth placed in compulsory institutional care.

DETAILED DESCRIPTION:
Substance abuse and criminality among youth in Sweden are urgent problems. More knowledge on effective interventions is crucial to help vulnerable youth at risk of developing an array of severe problems affecting both themselves, their relatives and society (Grahn, Lundgren Chassler & Padyab, 2015). Effective help for substance abuse increases chances to abandon criminality and build up a constructive life (Henderson et al, 2016, Chermack et al, 2010). Youth with severe substance abuse and psychosocial problems, such as criminal and socially disruptive behavior, often receive treatment in compulsory institutional care. The responsible party for delivering care in this domain is The Swedish National Board of Institutional Care, (Statens institutionsstyrelse, SiS). SiS provides institutional care on basis of the Swedish laws Care of Young Persons (Special Provisions) Act, LVU, Care of Substance Abusers (Special Provisions) Act, LVM, Secure Youth Care Act, LSU. Treatment is delivered in lockable institutions, situated in different locations around the country. However, the institutional setting differs from standard outpatient care where most substance use treatments have been designed for. For example, the locked ward and security routines pose challenges when fostering pro-social and constructive behavior (Gevers, Poelen, Scholte, Otten & Koordeman, 2020). Every activity must be thoroughly planned to lower risks of violence or escaping and routines, such as visitations, can lower the ability and motivation to engage in positive activities outside the institution (Brauers, Kroneman, Otten, Lindauer & Popma, 2016). The Swedish Agency for Health Technology Assessment and Assessment of Social Services, SBU, concluded in a systematic review (2016) that the scientific support for several of the treatment programs conducted at SiS are inadequate. Consequently, that more research on treatment in institutional care is needed, especially high-quality studies with a study design adjusted to the specific conditions prevailing there.

An empirically supported substance use treatment developed for youth ages twelve to twenty five is the Adolescent Community Reinforcement Approach, A-CRA. A-CRA promotes long-term abstinence, increase social stability and decrease depression and other co-morbid psychiatric problems according to a large number of studies since the nineteen seventies (Azrin, Sisson, Meyers, & Godley, 1982; Dennis et al., 2004; Hunt & Azrin, 1973; Godley et al., 2014; Godley et al., 2001; Godley, Smith, Passetti, & Subramaniam, 2014). A-CRA is recommended in national guidelines for the treatment of substance use disorder in adolescents (Socialstyrelsen, 2017). Treatment consists of eighteen procedures that aim to reduce problematic behaviors and increase constructive behaviors. Example of procedures are happiness scale and treatment goals, functional analysis of substance use behavior, increasing prosocial activities, drink/drug refusal, relapse prevention, communication skills, caregiver sessions, job seeking skills and anger management (Godley, Smith, Myers & Godley, 2016). Procedures are combined and tailored to youth individual goals and needs (Godley et al., 2016). A-CRA has also proven helpful for justice-involved youth with substance use disorder under probation (Henderson et al. 2016) and for homeless youth (Slesnick et al., 2007). However, as many other psychological treatments, A-CRA has mostly been delivered and evaluated within outpatient care. It is unclear whether A-CRA is as effective when delivered in compulsory care where many adolescents with severe substance use disorder and criminal behavior receive treatment.

The overall objective of this research project is to scientifically evaluate the effectiveness of A-CRA in compulsory institutional care for youth with substance use disorder and criminal behavior. In addition, to explore mechanisms of change, what mediates substance abuse and criminal behavior.

Youth are randomized to either treatment as usual or treatment as usual with the addition of A-CRA. Treatment as usual is defined as the interventions and treatments adolescents are usually offered and undergo in institutional care. These are Motivational Interviewing, MI, Cognitive Behavioral Therapy, CBT, Aggression Replacement Therapy, ART or Acceptance and Commitment Therapy, ACT. Randomization takes place at site level with even allocation to the groups. Quantitative measurements take place before, during and after treatment as well as follow-up at 1, 3, 6 and 12 months. Primary endpoint is 6 months after treatment completion. Qualitative data will be collected by interviewing participants at 3 month follow-up. Potential adverse events will be collected after treatment completion using open questions and registered when reported by staff in the research group or at KI.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-21
* Placed in institutional care
* Suffers from SUD and socially disruptive behaviour
* Ability to read and understand informed consent and interventions

Exclusion Criteria:

* Severe cognitive or psychiatric condition preventing the ability to provide informed consent or undergo assessment or interventions
* Serious somatic condition requiring acute medical attention

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Social, emotional and behavioural problems | 0 weeks, 7 weeks, 14 weeks and at follow-up 1, 3, 6, and 12 months after treatment completion
  Measured using the Strengths and Difficulties Questionnaire

SECONDARY OUTCOMES:
Self reported substance use | 0 weeks, 7 weeks, 14 weeks and at follow-up 1, 3, 6, 12 months after treatment
  Self-reported substance use, five questions
Use of alcohol | 0 weeks, 14 weeks and at follow-up 1, 6 and 12 months after treatment completio
  AUDIT - Alcohol Use Disorders Identification Test (Saunders et al, 1993)
Use of illegal drugs | 0 weeks, 14 weeks and at follow-up 1, 6 and 12 months after treatment completion
  Drug Use Disorders Identification Test (DUDIT; Berman, Bergman, Palmstierna, & Schlyter, 2005)
Number of days until the first relapse | 0 weeks, 7 weeks, 14 weeks and at follow-up 1, 3, 6 and 12 months after treatment completion
  Self-reported substance use, five questions
Aggressive behavior | 0 weeks, 7 weeks and 14 weeks and at follow-up 1 month after treatment completion
  Measured using the Bröset Violent Checklist (Koskela, 2012)
Goal directed behavior and values | 0 weeks, 7 weeks, 14 weeks and at follow-up 1, 3, 6, 12 months after treatment
  Bull's-Eye Values Survey (BEVS; Lundgren et al., 2012)
Psychological flexibility | 0 weeks, 7 weeks, 14 weeks and at follow-up 1, 3, 6, 12 months after treatment
  Avoidance and Fusion Questionnaire Short Version (AFQ-Y8; Livheim et al.,2016)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Lundgren, PhD, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Sundbo, Fagersta, Västmanland County
  - Fagersta, Lindome, Västra Götaland County
  - Statens institutionsstyrelse, SiS, Johannisberg, Kalix
  - Statens institutionsstyrelse, SiS, Ljungbacken, Uddevalla

IPD SHARING:
Plan to Share IPD: No